CLINICAL TRIAL: NCT00464308
Title: The Rabeprazole and Esomeprazole Reflux Assessment Trial (TREAT)
Brief Title: A Study to Compare the Number of Patients With Gastro-Oesophageal Reflux Disease (GORD) Achieving Heartburn and Regurgitation Symptom Resolution After Treatment With Either Rabeprazole Sodium 20mg, Esomeprazole 20mg or Esomeprazole 40mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR006397
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Gastro-oesophageal Reflux
Keywords: Gastroesophageal Reflux; Heartburn; Proton pump inhibitor; GORD
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole; Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Active Comparator): Esomeprazole 40mg once daily for 28days - 1 placebo tab/cap & 1 active tab/cap daily
  Interventions: Drug: Esomeprazole
- 002 (Active Comparator): Esomeprazole 20mg once daily for 28days - 1 placebo tab/cap & 1 active tab/cap daily
  Interventions: Drug: Esomeprazole
- 003 (Active Comparator): Rabeprazole 20mg once daily for 28days - 1 placebo tab/cap & 1 active tab/cap daily
  Interventions: Drug: Rabeprazole

INTERVENTIONS:
Drug: Esomeprazole — 20mg once daily for 28days - 1 placebo tab/cap & 1 active tab/cap daily
  Arms: 002
Drug: Rabeprazole — 20mg once daily for 28days - 1 placebo tab/cap & 1 active tab/cap daily
  Arms: 003
Drug: Esomeprazole — 40mg once daily for 28days - 1 placebo tab/cap & 1 active tab/cap daily
  Arms: 001

SUMMARY:
The primary objective of this study is to compare, the number of patients with heartburn and regurgitation symptom resolution after treatment with either rabeprazole 20 mg, esomeprazole 20 mg or esomeprazole 40 mg.

DETAILED DESCRIPTION:
The study is designed to be conducted in a realistic General Practice (GP) setting, enrolling typical Gastro-oesophageal Reflux Disease (GORD) patients that present for treatment, and for whom a Proton Pump Inhibitor (PPI) would normally be prescribed. The study will be conducted over a 4-week period on the basis that current GP standard practice is to treat the GORD patient for a period of 4-weeks prior to reassessment and further follow-up if required. This study is conducted in patients with GORD - associated heartburn (with or without regurgitation) at multiple GP centers, treatment is assigned based on chance (randomized), similar to the toss of a coin and neither doctor or patient knows which treatment they will receive (double-blinded). Following screening to determine eligibility, patients will be randomized to receive oral treatment with either, 20 mg rabeprazole, 20 mg esomeprazole or 40 mg esomeprazole once daily for 4 weeks. This 4-week study encompasses 2 protocol-mandated visits (baseline on day 0 and final visit on day 28). It is hypothesized that rabeprazole 20 mg will be no less effective than (non-inferior) esomeprazole 40 mg for the degree of GORD symptom resolution. Patients will take one tablet (rabeprazole 20 mg or placebo) and one capsule (esomeprazole 20 mg, esomeprazole 40 mg or placebo) each day for 28 days. The study medication will be taken once daily in the morning before breakfast, except the first dose, which will be taken during Visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Heartburn (defined as a feeling of burning or pain, rising from the epigastrium or lower part of the chest up towards the neck) with or without regurgitation
* Patients must have had episodes of heartburn with or without regurgitation for 3 months or longer, and for >= 3 days in the 7 days prior to randomisation
* Able to understand and complete questionnaires, able to give written informed consent, and have access to a telephone

Exclusion Criteria:

* Patients requiring endoscopy within 4 weeks of randomisation or with gastrointestinal symptoms that, in the opinion of the investigator, require further investigation prior to or coincident with initiation of PPI therapy which would include, but are not limited to, alarm symptoms such as unintentional weight loss, progressive difficulty swallowing (dysphagia), iron deficiency anaemia and epigastric mass
* Significant gastrointestinal obstruction, major gastric or oesophageal surgery (excluding appendectomy or cholecystectomy), oesophageal stricture or pyloric stenosis, extra-oesophageal manifestations of reflux disease
* Patients with Barrett's oesophagus (>3cm), Zollinger-Ellison Syndrome, scleroderma, malignancy (other than non-melanoma skin cancers) present within the last 5 years, hypersensitivity to rabeprazole or esomeprazole or any PPI, or any other significant condition that, in the opinion of the investigator, could interfere with the patients participation or compliance in the study such as past or current history of alcohol or drug abuse, hepatic, renal, pulmonary, respiratory abnormalities, or who have participated in an investigational drug or investigational device study within 30 days prior to the baseline visit or who are expected to do so during the 4 week study period
* Female patients who are currently pregnant or breast feeding, or who, in the opinion of the investigator, may become pregnant throughout the study
* Use of histamine-2 receptor antagonists (H2RAs) within 7 days of randomisation, anticholinergics, cholinergics, spasmolytics, opiates, sucralfate, proton pump inhibitors (PPIs), prokinetics, antibiotics (in relation to H. pylori treatment) or bismuth compounds within 14 days of randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1392 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd
Locations (25):
- Australia (25):
  - Belconnen
  - Bondi Junction
  - Brookvale
  - Browns Plains
  - Campbelltown
  - Campsie
  - Caringbah
  - Castle Hill
  - Charlestown
  - Dapto
  - Darlinghurst
  - Dubbo
  - Elizabeth
  - Fairfield
  - Hoppers Crossing
  - Ingleburn
  - Leichhardt
  - Maroubra
  - Melton
  - Mount Druitt
  - Oaklands Park
  - Royal Park
  - Sydney
  - Wentworthville
  - Wyoming

REFERENCES:
- [Derived] Biscola FT, Abe CM, Guth BE. Determination of adhesin gene sequences in, and biofilm formation by, O157 and non-O157 Shiga toxin-producing Escherichia coli strains isolated from different sources. Appl Environ Microbiol. 2011 Apr;77(7):2201-8. doi: 10.1128/AEM.01920-10. Epub 2011 Feb 11. PMID 21317257
- [Derived] Eggleston A, Katelaris PH, Nandurkar S, Thorpe P, Holtmann G; Treat Study Group. Clinical trial: the treatment of gastro-oesophageal reflux disease in primary care--prospective randomized comparison of rabeprazole 20 mg with esomeprazole 20 and 40 mg. Aliment Pharmacol Ther. 2009 May 1;29(9):967-78. doi: 10.1111/j.1365-2036.2009.03948.x. Epub 2009 Feb 3. PMID 19210493

RESULTS

PARTICIPANT FLOW:
Groups:
- Rabeprazole 20 mg/Day: Rabeprazole 20 mg once daily for 28 days - 1 placebo tablet/capsule plus 1 active tablet/capsule daily
- Esomeprazole 40 mg/Day: Esomeprazole 40 mg once daily for 28 days - 1 placebo tablet/capsule plus 1 active tablet/capsule daily
- Esomeprazole 20 mg/Day: Esomeprazole 20 mg once daily for 28 days - 1 placebo tablet/capsule plus 1 active tablet/capsule daily
Period: Overall Study
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Started | 464 | 469 | 459
Completed | 395 | 406 | 400
Not Completed | 69 | 63 | 59
Not completed — Adverse Event | 22 | 27 | 16
Not completed — Lost to Follow-up | 29 | 19 | 20
Not completed — Patient discontinued and other reasons | 17 | 17 | 23
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day | Total
Number analyzed (Participants) | 464 | 469 | 459 | 1392
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (14.8) | 48 (14.7) | 46.2 (14.8) | 46.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 208 | 208 | 620
  Male | 260 | 261 | 251 | 772
Region of Enrollment [Number; unit: participants]
  Australia | 464 | 469 | 459 | 1392

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Complete Resolution of Heartburn by Week 4
Description: Complete resolution is the absence of symptoms for any 7 consecutive days within the 4 week period assessed by the PAGI-SYM scale. This likert scale describes a series of symptoms as follows: 0-None, 1-Very Mild, 2-Mild, 3-Moderate, 4-Severe, 5 Very Severe.
Time Frame: week 4 of treatment
Population: The intent-to-treat (ITT) population was used for all efficacy analyses. The data were reanalysed using the compliance population (defined as all subjects who consumed at least 80% of study medication and who completed at least 80% of data recording).
Measure: Number; unit: participants
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Number analyzed (Participants) | 464 | 469 | 459
participants | 272 | 302 | 278
Statistical Analysis 1: Comparison: Rabeprazole 20 mg/Day vs Esomeprazole 40 mg/Day; Primary endpoints were assessed using non-inferiority tests. See below; Test type: Non-Inferiority or Equivalence — A sample size of 450 subjects per arm will give a 90% power (with a one-sided 95% confidence interval and a minimal clinically important difference of 9%) to demonstrate non-inferiority of rabeprazole 20mg to esomeprazole 40mg with respect to the number of patients with complete resolution of heartburn with or without regurgitation at week 4; p < 0.05, Non-inferiority — Adjustment for multiple comparisons was not made. The a priori threshold for statistical significance was p<0.05. Tests were 2-sided except for the non-inferiority test which was 1-sided; Proportion difference = -0.11 — Assumed that the true resolution rates in the rab20 and eso40 groups would be 30% (0.3). Non inferiority was considered proven if the lower confidence interval of the one sided 95% CI of P(rab20)-P(e40) was above -9%

2. Secondary Outcome: The Median Time to Complete Resolution of Heartburn Symptoms.
Time Frame: week 4 of treatment
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Number analyzed (Participants) | 464 | 469 | 459
days | 11 [9 to 15] | 9 [7 to 10] | 12 [10 to 15]

3. Secondary Outcome: The Median Time to Complete Relief of Regurgitation Symptoms
Time Frame: 4 weeks
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Number analyzed (Participants) | 464 | 469 | 459
days | 9 [7 to 12] | 11 [8 to 14] | 13 [10 to 15]

4. Primary Outcome: The Number of Patients Achieving Complete Resolution of Regurgitation Symptoms at Week 4
Description: Complete resolution is the absence of symptoms for any 7 consecutive days within the 4 week period assessed by the PAGI-SYM scale. This likert scale describes various symptoms as follows: 0-none, 1-Very Mild, 2-Mild, 3-Moderate, 4-Severe, 5-Very Severe.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Number analyzed (Participants) | 464 | 469 | 459
participants | 281 | 283 | 276
Statistical Analysis 1: Comparison: Rabeprazole 20 mg/Day vs Esomeprazole 40 mg/Day; Primary endpoints were assessed using non-inferiority tests. See below; Test type: Non-Inferiority or Equivalence — The sample size calculation was based upon the number of patients acheiveing complete resolution of HEARTBURN. A sample size of 450 subjects per arm will give a 90% power (with a one-sided 95% confidence interval and a minimal clinically important difference of 9%) to demonstrate non-inferiority of rabeprazole 20mg to esomeprazole 40mg with respect to the number of patients with complete resolution of heartburn with or without regurgitation at week 4; p < 0.05, non-inferiority — All statistical tests were interpreted at the 5% significance level (2-tailed); Proportion difference = -0.051 — Non inferiority was considered proven if the lower confidence interval of the one sided 95% CI of P(rab20)-P(e40) was above -9%

5. Primary Outcome: The Number of Patients Achieving Satisfactory Resolution of Heartburn by Week 4
Description: Satisfactory resolution, which is achieved if, on any 7 consecutive days within the 4 week period, the severity of symptoms never exceeds 'mild' (symptoms must be absent, very mild, or mild) assessed by the PAGI-SYM scale. This likert scale describes various symptoms as follows: 0-none, 1-Very Mild, 2-Mild, 3-Moderate, 4-Severe, 5-Very Severe.
Time Frame: 4 weeks
Population: Symptom scores 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, 5=very severe
Measure: Number; unit: participants
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Number analyzed (Participants) | 464 | 469 | 459
participants | 405 | 418 | 414
Statistical Analysis 1: Comparison: Rabeprazole 20 mg/Day vs Esomeprazole 40 mg/Day; Primary endpoints were assessed using non-inferiority tests. See below; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.05, non-inferiority — [p-value comment as in outcome 1, analysis 1]; Proportion difference = -0.053 — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: The Number of Patients Achieving Satisfactory Resolution of Regurgitation Symptoms by Week 4
Description: Satisfactory resolution, which is achieved if, on any 7 consecutive days within the 4 week period, the severity of symptoms never exceeds 'mild' (symptoms must be absent, very mild, or mild)assessed by the PAGI-SYM scale. This likert scale describes a series of symptoms as follows: 0-None, 1-Very Mild, 2-Mild, 3-Moderate, 4-Severe, 5 Very Severe.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Number analyzed (Participants) | 464 | 469 | 459
participants | 397 | 413 | 402
Statistical Analysis 1: Comparison: Rabeprazole 20 mg/Day vs Esomeprazole 40 mg/Day; Primary endpoints were assessed using non-inferiority tests. See below; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.05, non-inferiority — [p-value comment as in outcome 1, analysis 1]; Proportion difference = -0.061 — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: The Mean Percentage of Participants With 24-hour Heartburn Symptom Free Periods
Time Frame: 4 weeks
Measure: Mean (95% Confidence Interval); unit: percent of participants
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Number analyzed (Participants) | 464 | 469 | 459
percent of participants | 56.3 [53.1 to 59.5] | 63.4 [60.2 to 66.6] | 56.1 [52.9 to 59.3]

ADVERSE EVENTS:
Arm/Group | Rabeprazole 20 mg/Day | Esomeprazole 40 mg/Day | Esomeprazole 20 mg/Day
Serious Adverse Events (participants affected / at risk) | 5/464 | 1/469 | 9/459
Other Adverse Events (participants affected / at risk) | 151/464 | 155/469 | 158/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabeprazole 20 mg/Day (N=464) | Esomeprazole 40 mg/Day (N=469) | Esomeprazole 20 mg/Day (N=459)
meniscal tear of right knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
alleged assault (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
perianal abscess drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
multiple pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabeprazole 20 mg/Day (N=464) | Esomeprazole 40 mg/Day (N=469) | Esomeprazole 20 mg/Day (N=459)
Gastrointestinal motility and defaecation cond (Gastrointestinal disorders) | 24 (26) | 29 (32) | 36 (40)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 63 (86) | 67 (80) | 54 (77)
Salivary gland conditions (Gastrointestinal disorders) | 2 (4) | 8 (8) | 4 (7)
Infections - pathogen class unspecified (Infections and infestations) | 21 (22) | 9 (10) | 26 (29)
Viral infectious disorders (Infections and infestations) | 9 (9) | 6 (7) | 13 (13)
Other (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Joint disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8) | 3 (3)
Muscle disorders (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 4 (4)
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8) | 6 (7)
Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 19 (22) | 24 (30) | 31 (32)
Neurological disorders NEC (Nervous system disorders) | 9 (9) | 9 (10) | 11 (11)

LIMITATIONS AND CAVEATS:
The MCID of 7.5% was amended to 9% to maintain power with smaller sample size.The proportion of patients without heartburn symptoms at baseline was not evenly distributed between treatment arms. This was a significant predictor of symptom resolution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days